CLINICAL TRIAL: NCT03066687
Title: Randomized, Open-Label, 2-Way Crossover Study to Determine the Effect of Food on the Pharmacokinetics of Erdafitinib in Healthy Subjects
Brief Title: A Study to Determine the Effect of Food on the Pharmacokinetics of Erdafitinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108289; 42756493EDI1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1: Erdafitinib 9 mg (Experimental): Participants will receive 9 milligram (mg) dose of erdafitinib under fasted condition [Treatment A] in Period 1, and under fed (with high-fat and high-calorie breakfast) condition [Treatment B] in Period 2. Each Treatment Period will be separated by a washout of at least 28 days.
  Interventions: Drug: Erdafitinib
- Treatment Sequence 2: Erdafitinib 9 mg (Experimental): Participants will receive 9 mg dose of erdafitinib under fed (high-fat and high-calorie breakfast) condition [Treatment B] in Period 1, and under fasted condition [Treatment A] in Period 2. Each Treatment Period will be separated by a washout of at least 28 days.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Erdafitinib 9 mg (provided as one 4-mg tablet [G-024] and one 5-mg tablet [G-025]) will be administered orally on Day 1 in each Treatment Period of assigned sequence.

SUMMARY:
The primary purpose of this study is to evaluate the effect of food on the relative bioavailability of a single 9 milligram (mg) oral dose of erdafitinib in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* If a woman, must be not of childbearing potential: postmenopausal (greater than [>] 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 12 months and a serum follicle stimulating hormone [FSH] >40 International Units Per Liter [IU/L]); or surgically sterile
* If a woman, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and on Day -1 of Period 1 and Period 2
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after the last study drug administration
* Body mass index (BMI; weight [kg]/height^2 [m]^2) between 18 and 32 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than 50 kg
* Non-smoker for at least 6 months before first study drug administration

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History or current evidence of ophthalmic disorder, such as central serous retinopathy (CSR) or retinal vein occlusion, active wet age related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Clinically significant abnormal values for hematology, serum chemistry, or urinalysis at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at screening as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen and hormonal replacement therapy, within 14 days before the first dose of the study drug is scheduled until completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, and 366 hours post dose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, and 366 hours post dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, and 366 hours post dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Baseline, up to end of study (Day 15 of Period 2) or early withdrawal
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Lincoln, Nebraska, United States